CLINICAL TRIAL: NCT04269551
Title: A Multicenter, Phase 1b, Open Label, Nonrandomized, Single Dose Study Evaluating the Safety, Tolerability and Activity of BIVV020 in Adults With Cold Agglutinin Disease
Brief Title: A Safety and Tolerability Study of BIVV020 in Adults With Cold Agglutinin Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioverativ, a Sanofi company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDY16370; 2019-001844-22 (EudraCT Number); U1111-1233-0831 (Other: UTN)
Record Dates: First submitted 2020-01-29; First posted 2020-02-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Haemolytic Anaemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BIVV020 IV (Experimental): Single administration dose 1, plus two optional doses of BIVV020 administered intravenously.
  Interventions: Drug: BIVV020

INTERVENTIONS:
Drug: BIVV020 — Pharmaceutical form:solution for injection Route of administration: intravenous

SUMMARY:
Primary Objective:

To assess the safety and tolerability in participants with cold agglutinin disease (CAD), after a single dose of intravenous (IV) BIVV020

Secondary Objectives:

To assess, in participants with cold agglutinin disease, after a single dose of intravenous (IV) BIVV020:

* The effect of BIVV020 on complement mediated hemolysis
* The pharmacodynamics (PD) of BIVV020 relating to complement inhibition
* The pharmacokinetics (PK) of BIVV020
* The immunogenicity of BIVV020

DETAILED DESCRIPTION:
Up to 23 weeks (screening period up to 8 weeks, treatment period 15 weeks)

ELIGIBILITY:
Inclusion criteria :

* Male and/or female patients, ≥ 18 years of age with cold agglutinin disease as defined by:

  1. Chronic hemolysis per Investigator's judgement,
  2. Polyspecific direct antiglobulin test (DAT) positive,
  3. Monospecific DAT strongly positive for C3d,
  4. Cold agglutinin (CAg) titer ≥ 64 at 4 C; and,
  5. IgG DAT ≤1+.
* A hemoglobin level ≤11 mg/dL.
* A total bilirubin level above the normal reference range that is thought to be due to hemolysis.
* Documented vaccinations against encapsulated bacterial pathogens (Neisseria meningitidis, including serogroup B meningococcus and Streptococcus pneumoniae) within five years of screening or willing to complete protocol specified vaccinations.
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion criteria:

* Cold agglutinin syndrome secondary to infection, rheumatologic disease, or known high grade hematologic malignancy, or known solid organ tumor.
* Clinically relevant infection of any kind within one month preceding screening.
* Treatment with anti-CD20 monotherapy within three months or anti CD20 combination therapies within six months prior to screening.
* Concurrent treatment with systemic immunosuppressive agents targeting B- or T-cell function and/or cytotoxic agents within 3 months prior to screening. Concurrent treatment with other systemic immunosuppressants within 5.5 half-lives of the drug prior to screening.
* Any specific complement system inhibitor within three months prior to screening.
* Concurrent treatment with systemic corticosteroids other than a stable daily dose equivalent to ≤10 mg/day prednisone within three months prior to screening.
* If female, pregnant or lactating.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs) | Screening to Day 106
  Number of participants with adverse events (AEs)

SECONDARY OUTCOMES:
Mean change from baseline in bilirubin over time | Day 1 to Day 106
  Assessment of total bilirubin
Mean change from baseline in hemoglobin over time | Day 1 to Day 106
  Assessment of hemoglobin
Complement System Classical Pathway Levels as Measured by WIESLAB Assay | Day 1 to Day 106
  Inhibition by BIVV020 of the complement system classical pathway measured by the WIESLAB assay
Complement System Alternative Pathway Levels as Measured by WIESLAB Assay | Day 1 to Day 106
  Effect of BIVV0020 on the complement system alternative pathway measured by the WIESLAB assay
Total Complement (CH50) Levels | Day 1 to Day 106
  Complement CH50 is a blood test that helps us determine whether protein abnormalities and deficiencies in the complement system are responsible for any increase in autoimmune activity. It will be assessed using complement assays.
Total Complement Factor C4 Levels | Day 1 to Day 106
  Total C4 Levels will be assessed in plasma using complement assays
PK parameter: Cmax | Day 1 to Day 106
  Observed maximum plasma concentration
PK parameter: tmax | Day 1 to Day 106
  Observed first time to reach Cmax
PK parameter: AUClast | Day 1 to Day 106
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast
PK parameter: AUC0-∞ | Day 1 to Day 106
  Calculated area under the plasma concentration versus time curve extrapolated to infinity
Number of participants with anti-BIVV antibodies | Day 1 to Day 106
  Observed number of participants with BIVV020 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- United States (5):
  - Investigational Site Number :8400002, Fayetteville, Georgia
  - Investigational Site Number :8400009, St Louis, Missouri
  - Investigational Site Number :8400006, The Bronx, New York
  - Investigational Site Number :8400008, Pittsburgh, Pennsylvania
  - Investigational Site Number :8400004, Seattle, Washington
- Investigational Site Number :2760001, Essen, Germany
- Investigational Site Number :3800001, Milan, Milano, Italy
- Investigational Site Number :5280001, Amsterdam, Netherlands
- Investigational Site Number :5780001, Bergen, Norway
- Investigational Site Number :8260001, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] D'Sa S, Vos JMI, Barcellini W, Wardecki M, Perrin L, Barker G, Zilberstein M, Storek M, Chow T, Roth A. Safety, tolerability, and activity of the active C1s antibody riliprubart in cold agglutinin disease: a phase 1b study. Blood. 2024 Feb 22;143(8):713-720. doi: 10.1182/blood.2023022153. PMID 38085846
- See also: PDY16370 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25315&tenant=MT_SNY_9011